CLINICAL TRIAL: NCT04637061
Title: Rectal Cancer 4 Check Study
Brief Title: Rectal Cancer Anastomosis 4 Check Study
Acronym: REC4T
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 04101969
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; indocyanine green; fluorescence angiography; surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- REC4T study patients: Rectal adenocarcinoma or polyp with indication for resection and primary colo-rectal mechanical anastomosis using a circular stapler with/or without protective ostomy undergoing upfront surgery and patients undergoing neoadjuvant therapy followed by surgery (see Inclusion/Exclusion Criteria)
  Interventions: Combination Product: intraoperative near infrared (NIR) indocyanine green (ICG)-induced fluorescence angiography (FA) and air leak testing to assess the integrity and the perfusion levels of the colorectal anastomosis; Diagnostic Test: Air Leak test; Diagnostic Test: Evaluation of the anastomotic rings

INTERVENTIONS:
Combination Product: intraoperative near infrared (NIR) indocyanine green (ICG)-induced fluorescence angiography (FA) and air leak testing to assess the integrity and the perfusion levels of the colorectal anastomosis — Extra-luminal (serosa) and Endo-luminal (mucosal) evaluation of the proximal colon and distal rectal stump perfusion based on a semi-quantitative NIR-ICG-induced FA. This will be conducted administering IV a bolus of 3.75 to 7.5 mg of ICG and evaluated using a Fluorescence Imaging System; following after completion of the anastomosis a second bolos of 3.75 to 7.5 mg of ICG will be administered IV and the anastomosis will be visualized by insertion of the system trans-anally. Colon and rectal segments and quadrants will be scored for any defect of perfusion.
  Other Names: Near Infrared Fluorescence angiography; indocyanine green
Diagnostic Test: Air Leak test — This will be conducted insufflaying air in the anastomosis through a proctoscope, tube or a flexible endoscope, after filling of the pelvis with saline solution and luminal occlusion of the intestine proximal to the anastomosis. Also, the anastomosis will be checked transanally for the presence of air leak.
Diagnostic Test: Evaluation of the anastomotic rings — The assessment of the anastomotic rings following mechanical anastomosis will be recorded as complete/incomplete

SUMMARY:
Anastomotic failure (AF), including anastomotic leakage (AL), increases morbidity and mortality after colorectal cancer (CRC) resection. An inadequate perfusion of the anastomosis or technical stapling defects may contribute to AF. Several studies evaluated the singular use of intraoperative near infrared (NIR) indocyanine green (ICG)-induced fluorescence angiography (FA) and air leak testing to assess the integrity and the perfusion levels of the colorectal anastomosis. So far, a combined use of these methodologies, although acknowledged has not yet been tested as an indicator of postoperative AF or of intra-operative anastomotic repair in a prospective setting. This study aims to implement the intraoperative anastomotic assessment in a prospective series of patients undergoing rectal resection plus primary anastomosis for rectal cancer with or without ostomy, using a semi-quantitative check of 4 items (4-check). The procedure will include NIR-ICG-induced FA (to assess perfusion), air leak test and evaluation of the anastomotic donuts (to assess for the presence of technical defects). Included patients will be those scheduled for elective rectal resection with total or partial mesorectal excision and primary colo-rectal anastomosis with/or without protective ostomy. Primary outcomes will be the overall incidence of intra-operative anastomotic repair and the rate of post-operative AF. Secondary outcomes will be the overall incidence of adverse events and serious complications, the estimation of costs and resources, the operative time, hospitalization and post-operative measurement of inflammatory markers.

DETAILED DESCRIPTION:
All consecutive patients undergoing rectal resection (open and mini-invasive procedures) plus primary anastomosis for rectal cancer selected for the study will udergo a surgical intra-operative assessment of the anastomosis based on the check of the following 4 items (4-check):

1. Extra-luminal (serosa) evaluation of the proximal colon and distal rectal stump perfusion based on a semi-quantitative assessment of the near infrared (NIR) indocyanine green (ICG)-induced fluorescence angiography (FA).
2. Endo-luminal (mucosal) evaluation of the proximal colon and distal rectal stump perfusion based on a semi-quantitative assessment of the NIR-ICG-induced FA.
3. Air leak test (extra-luminal and reverse).
4. Assessment of the anastomotic donuts. aiming to test the efficacy of the procedure (overall incidence of intra-operative anastomosis repairs) and the overall incidence of anastomotic failure

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Rectal adenocarcinoma or benign polyp with indication for rectal resection with total or partial mesorectal excision and primary colo-rectal anastomosis with/or without protective ostomy.
* Patients undergoing upfront surgery and patients undergoing neoadjuvant therapy followed by surgery.
* Patients with adequate performance status (Eastern Cooperative Oncology Group Scale score of ≤2).
* Patient must sign the Informed Consent Form (ICF) before any study procedures and agrees to attend all study visits.
* Selection of the patient before inclusion.

Exclusion Criteria:

* • Patient pregnant or suspected pregnancy.

  * Patient with a comorbid illness or condition that would preclude the use of surgery.
  * Past medical history of Inflammatory Bowel Disease (IBD).
  * Synchronous cancers requiring extended sub-total or total colectomies.
  * Long lasting therapy with steroids to be continued in the peri-operative period (4 weeks previous and 4 weeks after surgery).
  * Use of antiplatelet drug (anti-aggregant) and/or oral anti-coagulant drug to be continued in the peri-operative period (1 week previous and 4 weeks after surgery).
  * Patients assessed as American Society of Anesthesiologists (ASA) physical status 4.
  * Patients with clinical stage of cT4b tumor after neoadjuvant theapy.
  * Metastatic disease (clinical Stage 4).
  * Patient undergoing emergency procedures.
  * Planned colonic surgery along with major concomitant procedures (i.e. liver resections, other intestinal resections).
  * Previous colon surgery (excluding appendectomy).
  * Non-restorative procedures (i.e. Miles or Hartman resection).
  * Colo-anal manual anastomosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selected patients will receive oral bowel preparation as for colonoscopy, 2 days before surgery and managed with ERAS protocol. Patients should be treated with rectal resection with TME or PME and mechanical anastomosis with a circular stapler, using one of the following approaches:
  1. Open surgery.
  2. Laparoscopic surgery (operations performed through small incisions and ports placements independently from the type and length of incision for specimen extraction).
  3. Robot-assisted surgery (using robotic systems to aid in surgical procedures independently from the type and length of incision for specimen extraction).
  4. TaTME. Mini-invasive bottom up approach for mesorectal dissection and colorectal anastomosis using a single/double team, independently from the type and length of incision for specimen extraction.
  The following procedures is required during surgery:
  Routine splenic flexure mobilization.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
intra-operative anastomosis repairs | 01/01/2021 to 31/12/2022
  defined as additional suturing or re-do anastomosis
Rate of 30 day-anastomotic failure (AF) | 01/01/2021 to 31/12/2022
  defined as anastomotic-related morbidity, including anastomotic leakage, pelvic abscess, anastomotic-related fistula, sinus, and anastomotic stricture

SECONDARY OUTCOMES:
Rate of of adverse events | 01/01/2021 to 31/12/2022
  any medical or surgical complications
Rate of 30-day major complications | 01/01/2021 to 31/12/2022
  Clavien-Dindo grade IIIb-IV
Measure of costs | 01/01/2021 to 31/12/2022
  Costs resource utilization for the procedure
Medan length of post-operative stay | 01/01/2021 to 31/12/2022
  post-operative stay (measured in days)
C-Reactive Protein (CRP) measurement | 01/01/2021 to 31/12/2022
  measurement conducted in postoperative days 1, 3 & 5 (optional) using mg/L
Procalcitonin (PCT) measurement | 01/01/2021 to 31/12/2022
  measurement conducted in postoperative days 1, 3 & 5 (optional) using mg/L ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Persiani, MD, Principal Investigator — Fondazione Policlinico Universitarioa A Gemelli IRCCS

IPD SHARING:
Plan to Share IPD: No